CLINICAL TRIAL: NCT00903214
Title: Metabotropic Glutamate Receptor-1 (mGluR1): Validation of a Serendipitously Discovered Molecular Target for Breast Cancer Treatment
Brief Title: Riluzole in Women With Stage I, Stage II, or Stage IIIA Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding ended
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000641180; P30CA022453 (NIH); WSU-2008-120
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Riluzole; Amplified Fragment Length Polymorphism Analysis; Biopsy, Needle; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: riluzole — 100 mg orally twice a day, tablets self-administered, administered from day -14 to day 0 (scheduled surgery and preserve tissue for biormarker analysis)
  Other Names: RILUTEK
Genetic: polymorphism analysis — Pre-treatment, day -15 but may be done any time after enrollment but before surgery.
Procedure: axillary lymph node biopsy
Procedure: digital image analysis
Procedure: needle biopsy
Procedure: sentinel lymph node biopsy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood from patients with cancer in the laboratory may help doctors identify biomarkers related to cancer. Riluzole may help slow the growth of tumor cells.

PURPOSE: This phase I trial is studying riluzole in women with stage I, stage II, or stage IIIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the effects of glutamate receptor blockade with riluzole on cellular pathways important in the genesis and progression of disease in women with stage I-IIIA breast cancer by examining components of the mGluR1 signaling pathway in the pre- and post-treatment tumor samples to determine if glutamate blockade affects signaling through this pathway.

Secondary

* To determine whether treatment with riluzole affects the proliferation and apoptosis in a manner suggesting a potential for therapeutic effectiveness.
* To determine whether treatment with riluzole causes objectively measurable tumor shrinkage.

OUTLINE: Patients receive oral riluzole twice daily on days -14 to 0. Approximately 12 hours after completion of riluzole therapy patients undergo standard surgery (i.e., partial or total mastectomy) along with sentinel lymph node biopsy (for patients with node-negative disease) or full axillary dissection (for patients with node-positive disease) on day 0.

Patients undergo 3-dimensional image assessment at pre- and post-treatment by Computerized Ultrasound Risk Evaluation (C.U.R.E.).

Patients undergo core needle biopsy at baseline and during surgery for biomarker analysis (e.g., mGluR1) by IHC, western blotting, and RT-PCR. Blood samples are collected for GRM1 polymorphism analysis.

After completion of study treatment, patients are followed every 6 months for 1 year and then according to standard-of-care thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of adenocarcinoma of the breast

  * Stage I (T1c)-IIIA disease meeting the following criteria:

    * Large enough (> 1 cm) to undergo additional multiple core needle biopsies preoperatively
    * Surgically resectable for cure or palliation without first requiring neoadjuvant chemotherapy
* Patients who have previously been treated for breast cancer, but are judged to have developed a new primary cancer, rather than a recurrence, are eligible

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* ANC ≥ 1,000/mm³
* Platelet count ≥ 50,000/mm³
* Liver function tests ≤ 3 times upper limit of normal (ULN)
* Total bilirubin ≤ 2 times ULN
* Creatinine ≤ 1.5 mg/dL
* INR ≤ 25% normal limits
* Not pregnant or nursing
* No known history of HIV or AIDS
* No known history of hepatitis B or C
* No history of vertigo or Ménière's type of disorder
* No history of allergic reaction to riluzole or similar compounds

PRIOR CONCURRENT THERAPY:

* No prior estrogen blockers, chemotherapy, radiotherapy, biological therapy, or surgery for the treatment of breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Inhibition of downstream targets of the mGluR1 signaling cascade, specifically downregulation of PLCβ activity | Pre and Post-treatment with RILUTEK® (riluzole) administration
Downregulation of phosphorylated ERK1/2 | Pre and Post treatment with RILUTEK® (riluzole) administration:

SECONDARY OUTCOMES:
Measures of proliferation, specifically mitotic rate and expression of Ki-67 | Pre and Post treatment with RILUTEK® (riluzole) administration:
Measures of apoptosis, specifically levels of poly(ADP-ribose) polymerase (PAPR) cleavage and caspase III activity | Pre and Post treatment with RILUTEK® (riluzole) administration:

CONTACTS AND LOCATIONS:
Overall Officials: David H. Gorski, MD, PhD, FACSw, Principal Investigator — Barbara Ann Karmanos Cancer Institute